CLINICAL TRIAL: NCT07218653
Title: Sex-Specific Cerebrovascular Dysfunction in Metabolic Syndrome-Role of COX
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: R01 MetSyn; pending (Other Grant/Funding Number: NIH); School of Educ / Kinesiology (Other: UW Madison)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Metabolic Syndrome
Keywords: Cerebral Blood Flow; CBF; COX; Metabolic Syndrome; MetSyn
MeSH Terms: conditions — Metabolic Syndrome | interventions — Indomethacin; Lactose; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Participants are randomized to Placebo vs Indomethacin for 2 MRI visits such that they are their own control.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy controls (Experimental): Male and female participants 18-45 without Metabolic Syndrome. On study for 3 visits (up to 6 months). Randomized to either Placebo then Indomethacin or Indomethacin then Placebo for 2 MRI visits.
  Interventions: Drug: Indomethacin; Drug: Placebo; Diagnostic Test: MRI
- Metabolic Syndrome (Experimental): Male and female participants, age-matched with Healthy Controls, who have at least 3 defining symptoms of Metabolic Syndrome. Randomized to either Placebo then Indomethacin or Indomethacin then Placebo for 2 MRI visits.
  Interventions: Drug: Indomethacin; Drug: Placebo; Diagnostic Test: MRI

INTERVENTIONS:
Drug: Indomethacin — Indomethacin is a nonsteroidal anti-inflammatory. It prevents the production of prostaglandins, endogenous signaling molecules known to cause symptoms from inflammation.
  Indomethacin (1.5 mg/kg) will be taken orally prior to one MRI study visit.
  Other Names: Indo
Drug: Placebo — Participants will be screened for lactose intolerance. Total dosing will be calculated to match the mg needed for the indomethacin study visit.
  Other Names: Lactose
Diagnostic Test: MRI — CBF testing will be performed on 3T MRI scanners (GE Healthcare)
  Other Names: Magnetic Resonance Imaging

SUMMARY:
This study tests the hypothesis that Metabolic Syndrome (MetSyn) decreases cerebral blood flow (CBF) more in females than males due in part to the sex-specific loss of COX vasodilation. Male and female participants will be enrolled in two groups: Health Controls versus participants with MetSyn.

DETAILED DESCRIPTION:
The central hypothesis is that MetSyn decreases CBF more in females than males due in part to the sex-specific loss of COX vasodilation. This hypothesis is based on extensive preliminary data demonstrating MetSyn induces: 1) 3-fold larger reductions in CBF in females that abolish sex differences, 2) region-specific CBF reduction patterns, and 3) a greater loss of COX-mediated vasodilation in females.

This hypothesis is tested via three Specific Aims:

* Aim 1: Determine the extent of sex differences in MetSyn-driven CBF reductions. The investigators hypothesize females with MetSyn will demonstrate larger decrements in global, grey matter and white matter CBF versus males.
* Aim 2: Determine the sex-by-region interactions of MetSyn reductions in CBF. The investigators hypothesize females will demonstrate larger regional CBF declines-particularly in regions known to be impacted very early in brain pathologies and/or specifically impaired by insulin resistance.
* Aim 3: Determine the role of COX signaling in mediating CBF changes in MetSyn. The investigators hypothesize COX vasodilation is reduced more in females than males with MetSyn.

All consented participants will conduct a screening visit with a blood panel to identify control vs MetSyn eligibility.

Once eligible, participants complete three laboratory visits (each lasting about 2 hours):

1. Exercise Visit: VO2 Max, DEXA for adiposity quantification, NIH Toolbox to assess neurocognitive function
2. MRI Visit 1: blinded to either Placebo or Indomethacin
3. MRI Visit 2: blinded to either Placebo or Indomethacin

ELIGIBILITY:
Inclusion Criteria (Healthy Controls):

* non-hypertensive (less than 130/80 mmHg)
* non-obese with a Body Mass Index (BMI) less than 30 kilogram per meter squared (kg/m2)
* Normal blood glucose less than 100 grams per deciliter (g/dl)
* Normal lipids; LDL cholesterol less than130 milligrams per deciliter (mg/dl), triglycerides less than 150 mg/dl.
* Women must have a predictable menstrual cycle for MRI scheduling. Females will be studied on cycle days 1-7 (as presented in all preliminary data) to minimize sex hormone differences and their potential confounding effects on vascular outcomes. Oral contraceptives will be allowed in women to increase translatability in findings.

Inclusion Criteria (Participants with Metabolic Syndrome):

* Meet age criteria plus three or more of the five criteria for MetSyn as defined by ATP, the most common three factors meeting MetSyn criteria will be obesity, prehypertension / hypertension, and low HDL cholesterol.

Exclusion Criteria:

* Subjects with a diagnostic history of:

  * peripheral vascular, hepatic, renal, or hematologic disease
  * stroke
  * type 1 or 2 diabetes
  * sleep apnea
  * hypertension (allowed in MetSyn)
  * regular tobacco users
  * taking cardiovascular medications (e.g., statins, angiotensin II receptor blockers) or metabolic medications (metformin, insulin, semaglutide) or NSAID sensitivity will be excluded.
* In women: pregnancy or polycystic ovarian syndrome (PCOS, to avoid altered testosterone in women).
* A history of a neurocognitive disorder or an intellectual disability will be excluded from the study. A neurocognitive screener (MoCA) will be completed; a score below the normal range (25 or below) is exclusionary. Participants will complete the Patient Health Questionnaire-9 (PHQ-9) and General Anxiety Disorder-7 (GAD-7) to screen for symptoms of depression and anxiety to increase the translatability of data; normal to mildly elevated range (0-9) are included but excluded at higher scores (10-27).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Cerebral Blood Flow | data collected over 2 study visits that must be completed within 6 months
  Data collected via MRI under one of 2 conditions: placebo or indomethacin.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness: VO2 max | data collected at one study visit (must be completed within 6 months)
  Graded exercise test to assess maximal aerobic capacity, reported as VO2 max (milliliters of oxygen consumed per kilogram of body weight per minute)
Body Fat Mass | data collected at one study visit (must be completed within 6 months)
  Dual-energy x-ray absorptiometry (DEXA) to measure fat mass.
Cognitive Testing: Flanker Inhibitory Control and Attention | data collected at one study visit (must be completed within 6 months)
  NIH Toolbox to assess neurocognitive function. The Flanker test is a measure of executive function and is scored using a T-score where 100 is the average, higher scores indicate better performance.
Cognitive Testing: Pattern Comparison Processing Speed Test | data collected at one study visit (must be completed within 6 months)
  NIH Toolbox to assess neurocognitive function. The Pattern Comparison Processing Speed Test measures how many correct responses the participant has within 90 seconds. There is a maximum of 130 items.
Cognitive Testing: List Sorting Working Memory Test | data collected at one study visit (must be completed within 6 months)
  NIH Toolbox to assess neurocognitive function. The List Sorting Working Memory Test is a measure of recall and sorting. Participants scores reflect the number of items recalled and appropriately sorted up to 28 items maximum.
Cognitive Testing: Dimensional Change Card Sort Test | data collected at one study visit (must be completed within 6 months)
  NIH Toolbox to assess neurocognitive function. The Dimensional Change Card Sort Test measures accuracy: the number of accurate responses, up to a maximum of 40.
Cognitive Testing: Picture Vocabulary Test | data collected at one study visit (must be completed within 6 months)
  NIH Toolbox to assess neurocognitive function. The Picture Vocabulary Test has the participant hear a word and then pick from one of four pictures that best represents the word. It is scored using a T-score where 100 is the average, higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: William Schrage, PhD, Principal Investigator — UW Madison

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF